CLINICAL TRIAL: NCT02465957
Title: Phase 2 Study of aNK (Activated NK-92 Natural Killer Cells) Infusions in Combination With ALT-803 (IL-15) in Patients With Stage III (IIIB) or Stage IV Merkel Cell Carcinoma (MCC)
Brief Title: QUILT-3.009: Patients With Stage III (IIIB) or Stage (IV) Merkel Cell Carcinoma (MCC)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: ImmunityBio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: QUILT-3.009; MCC-001 (Other: NantKwest, Inc.)
Record Dates: First submitted 2015-06-03; First posted 2015-06-09 (Estimated); Results first posted 2024-05-02 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2020-08

CONDITIONS: Stage IIIB Merkel Cell Carcinoma; Stage IV Merkel Cell Carcinoma
Keywords: Merkel Cell Carcinoma; Neukoplast; NK-92; Natural Killer Cell; MCC; aNK
MeSH Terms: conditions — Carcinoma, Merkel Cell | interventions — ALT-803

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- aNK (NK-92) (Experimental): aNK (activated NK-92, formerly Neukoplast)
  Interventions: Biological: aNK (NK-92)
- aNK (NK-92) + N-803 (Experimental): aNK (activated NK-92, formerly Neukoplast) and N-803
  Interventions: Biological: aNK (NK-92) + N-803

INTERVENTIONS:
Biological: aNK (NK-92) — A natural killer cell line recovered from a patient with large granular lymphoma
  Other Names: NK-92, Neukoplast
  Arms: aNK (NK-92)
Biological: aNK (NK-92) + N-803 — aNK - A natural killer cell line recovered from a patient with large granular lymphoma and N-803 - Recombinant human super agonist interleukin-15 (IL-15) complex
  Arms: aNK (NK-92) + N-803

SUMMARY:
Phase II study to determine the effects of aNK infusions in combination with ALT-803 in patients with stage III (IIIB) or stage (IV) merkel cell carcinoma (MCC).

DETAILED DESCRIPTION:
This is a multi-center, non-randomized, open-label, phase 2 trial to determine the effects of aNK in combination with ALT-803 in patients with stage III (IIIB) or stage IV MCC. The study will use an adaptive Simon optimal two-stage design, which detects efficacy signals, allows for early assessment, and avoids enrolling larger numbers of patients in case of inefficacy.

In the original protocol, an initial cohort of up to 12 patients with stage III (IIIB) or stage IV MCC were to be enrolled and treated with aNK monotherapy (first stage). If the treatment in the first stage improved the 4-month progression free survival (PFS) rate from 4% to 20% (e.g. at least 1 patient out of 12 patients has PFS ≥ 16 weeks [4 months]), then the study would proceed to the second stage, in which 12 more patients were planned to be enrolled and treated. As of July 2016, the trial has met the required efficacy signal defined for the first stage and will continue to enroll a planned total of 24 patients who will receive the combination of aNK and ALT-803. Any patients who are already receiving aNK cells as monotherapy will receive aNK cells in combination with ALT-803 in subsequent cycles.

aNK will be given via IV infusion at a dose of 2 x 10^9 cells/m^2 on two consecutive days (= 1 cycle) every 2 weeks. In addition, ALT-803 will be administered SC at 10 μg/kg on the first day of every aNK infusion (before the aNK infusion) every 2 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients 18 years of age or older.
2. Patients must have histologically confirmed MCC that is Stage III (IIIB) or Stage IV, as defined by the 2010 AJCC staging criteria for MCC. MCC of unknown primary is allowed.
3. Prior systemic cytotoxic chemotherapies and/or novel immunotherapy treatments for MCC are allowed. A wash-out period of 2 weeks prior to aNK treatment will be required.
4. ECOG performance status of 0-2.
5. Voluntary written informed consent must be given before performance of any study-related procedure not part of normal medical care, with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care.
6. Mandatory diagnostic biopsy and whole blood sample are required. The tumor biopsy tissue will be analyzed for the presence of immune cells and will also undergo genomic, transcriptomic, and proteomic profiling.

Exclusion Criteria:

1. Major surgery within 30 days before study entry.
2. Any of the following clinical laboratory values at the time of enrollment:

   1. Absolute neutrophil count (ANC) < 1,000 cells/mm^3.
   2. Platelets < 50,000 x 10^9/L.
3. Liver function abnormalities as indicated by ongoing hepatic enzyme elevation (e.g. AST, ALT, GGT) > 2 x the ULN. Elevation related to direct tumor infiltration is allowed.
4. Renal insufficiency as indicated by a creatinine level > 2 x the ULN.
5. Myocardial infarction within 6 months prior to enrollment or New York Hospital Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled arrhythmias, or electrocardiographic evidence of acute ischemia or significant conduction system abnormalities in the opinion of the Investigator. Prior to study entry any known abnormality on an electrocardiogram (ECG) must be determined and documented by the Investigator to be not clinically significant to the patient participation in this study.
6. Any condition, including laboratory abnormalities, that in the opinion of the Investigator places the patient at unacceptable risk if he/she were to participate in the study. This includes, but is not limited to, serious medical conditions or psychiatric illness likely to interfere with participation in this clinical study.
7. Female patients who are pregnant or breastfeeding. Female patients of childbearing potential must have a negative pregnancy test and agree to use adequate contraception for the duration of the trial.
8. Patients with other malignancies or brain metastasis are not eligible; however, given the frequent coexistence of MCC with other malignancies, the following exceptions are allowed:

   1. Patients who have been continuously disease-free for any solid tumor malignancy >3 years prior to the time of enrollment.
   2. Patients with basal cell carcinoma or squamous cell carcinoma.
   3. Patients with prior history of in situ cancer (e.g., breast, melanoma, squamous cells carcinoma of the skin, cervical).
   4. Patients with prior history of prostate cancer that is not under active systemic treatment (except hormonal therapy), but with undetectable PSA (<0.2 ng/mL).
   5. Patients with chronic non-T-cell-based lymphocytic leukemia are eligible if they have isolated lymphocytosis (Rai stage O) on the condition that they do not require systemic treatment for their disease ["B" symptoms, Richter's transformation, lymphocyte doubling time (<6 months) and they do not have lymphadenopathy of hepatosplenomegaly].
   6. Patients with non-T-cell-based lymphoma of any type or hairy cell leukemia are eligible on the condition that they do not receive active systemic treatment for their hematologic disease and are in complete remission as evidenced by PET/CT scans and bone marrow biopsies for at least 3 months.
9. Patients on immunosuppressants, systemic corticosteroids, or any other investigational product.
10. Patients unwilling to consent to analysis of their tumor tissue.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2015-09-24 (Actual); Primary Completion 2018-03-19 (Actual); Study Completion 2018-03-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Robert H. Lurie Comprehensive Cancer Center, Chicago, Illinois
  - UPMC Cancer Center, Pittsburgh, Pennsylvania
  - Seattle Cancer Care Alliance, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- aNK (NK-92): aNK was to be given via IV infusion at a dose of 2 x 10^9 cells/m2 on two consecutive days (= 1 cycle) every 4 weeks for a total of 8 infusions (2 each/cycle) for a total of 4 treatment cycles.
- aNK (NK-92) + N-803: aNK was to be given via IV infusion at a dose of 2 x 10^9 cells/m2 on two consecutive days (= 1 cycle) every 2 weeks.
  N-803 was to be administered SC at 10 μg/kg on the first day of every aNK infusion (before the aNK infusion) every 2 weeks.
  Treatment was permitted to continue until a complete response was achieved or it was deemed appropriate by the Investigator and/or Sponsor Medical Monitor.
Period: Overall Study
Arm/Group | aNK (NK-92) | aNK (NK-92) + N-803
Started | 3 | 4
Completed | 3 (Completed defined as receiving at least one dose of study drug.) | 4 (Completed defined as receiving at least one dose of study drug.)
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- aNK (NK-92) + N-803: aNK (activated NK-92, formerly Neukoplast) N-803
  aNK (NK-92) + N-803: aNK - A natural killer cell line recovered from a patient with large granular lymphoma N-803 - Recombinant human super agonist interleukin-15 (IL-15) complex
- Total: Total of all reporting groups
Arm/Group | aNK (NK-92) | aNK (NK-92) + N-803 | Total
Number analyzed (Participants) | 3 | 4 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 77.3 (3.21) | 61.3 (1.26) | 68.1 (8.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 3 | 3 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 4 | 7
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 3 | 4 | 7
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Histology of Primary Diagnosis [Count of Participants; unit: Participants]
  Carcinoma/Adenocarcinoma | 0 | 1 | 1
  Neuroendocrine | 0 | 2 | 2
  Merkel Cell Carcinoma | 0 | 1 | 1
  Unknown | 3 | 0 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Progression Free Survival Rate at 4 Months
Time Frame: 4 months
Measure: Count of Participants; unit: Participants
Groups:
- aNK (NK-92) + N-803: aNK (NK-92): A natural killer cell line recovered from a patient with large granular lymphoma
  N-803: Recombinant human super agonist interleukin-15 (IL-15) complex
Arm/Group | aNK (NK-92) | aNK (NK-92) + N-803
Number analyzed (Participants) | 3 | 4
Participants | 3 | 3

ADVERSE EVENTS:
Time Frame: 30 days past treatment completion, up to 5 months
Arm/Group | aNK (NK-92) | aNK (NK-92) + N-803
All-Cause Mortality (participants affected / at risk) | 1/3 | 1/4
Serious Adverse Events (participants affected / at risk) | 0/3 | 2/4
Other Adverse Events (participants affected / at risk) | 2/3 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | aNK (NK-92) (N=3) | aNK (NK-92) + N-803 (N=4)
Oedema peripheral (General disorders) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 1
Ureteric compression (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | aNK (NK-92) (N=3) | aNK (NK-92) + N-803 (N=4)
Sinus bradycardia (Cardiac disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 1 | 1
Eye swelling (Eye disorders) | 0 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2
Chest discomfort (General disorders) | 0 | 1
Chills (General disorders) | 2 | 3
Fatigue (General disorders) | 1 | 1
Flushing (General disorders) | 0 | 1
Injection site erythema (General disorders) | 0 | 3
Injection site irritation (General disorders) | 0 | 1
Injection site rash (General disorders) | 0 | 1
Injection site reaction (General disorders) | 0 | 2
Night sweats (General disorders) | 0 | 1
Oedema peripheral (General disorders) | 0 | 1
Peripheral swelling (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 2
Temperature intolerance (General disorders) | 1 | 0
Localised infection (Infections and infestations) | 0 | 1
Oral candidiasis (Infections and infestations) | 0 | 1
Pharyngitis streptococcal (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Lymphocyte count (Investigations) | 0 | 1
Platelet count decreased (Investigations) | 0 | 1
Weight decreased (Investigations) | 0 | 1
Weight increased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 2
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Gout (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Limb mass (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Encephalopathy (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 1 | 0
Somnolence (Nervous system disorders) | 0 | 1
Delirium (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Restlessness (Psychiatric disorders) | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 1
Ureteric compression (Renal and urinary disorders) | 0 | 1
Ureteric obstruction (Renal and urinary disorders) | 0 | 1
Urinary tract stoma complication (Renal and urinary disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Vitiligo (Skin and subcutaneous tissue disorders) | 1 | 0
Hypotension (Vascular disorders) | 0 | 2

LIMITATIONS AND CAVEATS:
There is an insufficient number of subjects enrolled in order to evaluate efficacy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-08): https://cdn.clinicaltrials.gov/large-docs/57/NCT02465957/Prot_SAP_000.pdf